CLINICAL TRIAL: NCT02864290
Title: A Phase 1 Study Evaluating Safety, Tolerability, and Pharmacokinetics of Escalating Doses of ASP1235 (AGS62P1) Given as Monotherapy in Subjects With Acute Myeloid Leukemia (AML)
Brief Title: A Study to Evaluate Escalating Doses of ASP1235 (AGS62P1) Given as Monotherapy in Subjects With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to lack of efficacy.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1235-CL-0101; AGS62P1-16-1 (Other: Astellas Pharma Global Development, Inc.)
Record Dates: First submitted 2016-06-30; First posted 2016-08-12 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Pharmacokinetics of ASP1235 (AGS62P1); ASP1235; Acute Myeloid Leukemia; ASP1235 (AGS62P1)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation of ASP1235 (AGS62P1) Schedule A (Experimental): Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion once every three weeks (Q3W) to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose. A cycle is 21 days.
  Interventions: Drug: ASP1235
- Dose Escalation of ASP1235 (AGS62P1) Schedule B (Experimental): Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion every other week of a 4-week cycle (Q2W) to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose. A cycle is 28 days.
  Interventions: Drug: ASP1235
- Dose Expansion of ASP1235 (AGS62P1) Schedule A (Experimental): Once the maximum tolerated dose (MTD) or recommended Phase 2 dose has been determined, an expansion cohort of up to 25 subjects may be enrolled. Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion once every three weeks (Q3W).
  Interventions: Drug: ASP1235
- Dose Expansion of ASP1235 (AGS62P1) Schedule B (Experimental): Once the maximum tolerated dose (MTD) or recommended Phase 2 dose has been determined, an expansion cohort of up to 25 subjects may be enrolled. Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion every other week of a 4-week cycle (Q2W).
  Interventions: Drug: ASP1235
- Dose Escalation of ASP1235 (AGS62P1) Schedule C (Experimental): Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion once weekly for three weeks of a 4-week cycle to determine the MTD or recommended Phase 2 dose. A cycle is 28 days.
  Interventions: Drug: ASP1235
- Dose Expansion of ASP1235 (AGS62P1) Schedule C (Experimental): Once the MTD or recommended Phase 2 dose has been determined, an expansion cohort of up to 25 subjects may be enrolled. Subjects will receive ASP1235 (AGS62P1) as an intravenous infusion once weekly for three weeks pf a 4-week cycle.
  Interventions: Drug: ASP1235

INTERVENTIONS:
Drug: ASP1235 — intravenous (IV) infusion
  Other Names: AGS62P1

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ASP1235 (AGS62P1) given at three dosing schedules (Schedule A, every three weeks [Q3W] or Schedule B, every other week of a 4 week cycle [Q2W] or Schedule C once a week for 3 weeks of a 4 week cycle) in subjects with acute myeloid leukemia (AML) and determine the maximum tolerated dose (MTD). In addition, this study will assess the pharmacokinetics (PK), the immunogenicity and the anti-leukemic activity of ASP1235 (AGS62P1).

ELIGIBILITY:
Inclusion Criteria:

* Subject has morphologically documented primary or secondary AML by the World Health Organization (WHO) criteria (2008) which is relapsed or refractory after failing at least 1 regimen and is not a candidate for established salvage treatment regimens. For expansion cohorts, patients are eligible if they have had ≤ 3 prior lines of therapy. Lines of therapy include initial induction (up to 2 cycles) with consolidation/maintenance, if applicable, and subsequent salvage regimens. Consolidation alone and stem cell transplantation are not counted as lines of therapy.
* Subject has an Eastern Cooperative Oncology Group performance score (ECOG) ≤ 2
* Subject has adequate renal function with an estimated creatinine clearance of ≥ 30 mL/min by the Cockcroft-Gault equation adjusted for body weight
* Subject has a total bilirubin ≤ 1.5 x upper limit of normal (ULN), albumin ≥ 2.5 g/d, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Subjects must be competent to comprehend, provide written informed consent, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form
* A female subject is eligible to participate if she is not pregnant and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* A male subject with female partner(s) of child-bearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* A male subject must not donate sperm during the treatment period and for at least 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study drug administration.

Exclusion Criteria:

* Subject has a diagnosis of acute promyelocytic leukemia (APL)
* Subject has preexisting sensory or motor neuropathy Grade ≥ 2 at baseline
* Subject has received small molecule therapy, radiotherapy, immunotherapy, monoclonal antibodies, investigational drug, or chemotherapy within 14 days before first dose of study drug, with the exception of hydroxyurea
* Subject has any Grade ≥ 2 persistent non-hematological toxicity related to allotransplant
* Subject with Graft vs. Host Disease (GVHD) who is receiving treatment with systemic glucocorticoids > 10 mg/day equivalent of prednisone; however, treatment with low dose glucocorticoids (≤ 10 mg/day equivalent of prednisone) is permitted

  * The use of systemic glucocorticoids in excess of 10 mg/day equivalent of prednisone is permitted provided it is not for the treatment of GVHD (e.g. chronic obstructive pulmonary disease, anti-emetic, infusion reactions). The chronic use of topical, inhaled, and locally injected steroids is permitted
* Subject has known current central nervous system (CNS) disease
* Active angina or Class III or IV Congestive Heart Failure (CHF) (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of the first dose of study drug, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by medication
* Subject has clinical evidence of Disseminated Intravascular Coagulation
* Subject has known positivity for human immunodeficiency virus
* Subject has known active hepatitis B (positive hepatitis B surface antigen [HBs Ag]) or C infection. For subjects who are negative for HBs Ag, but hepatitis B core antibody (HBc Ab) positive, an HB deoxyribonucleic acid (DNA) test will be performed and if positive, the subject will be excluded. Subjects with positive serology but negative hepatitis C virus (HCV) ribonucleic acid (RNA) test results are eligible.
* Subject has an uncontrolled active infection requiring treatment and grade 3 or higher fever 48 hours before the first dose of study drug. Controlled infections (i.e. 3 negative cultures completing antibiotics and/or stable fungal infection in therapy) are allowed provided the subject has a temperature of < 38.3°C within 48 hours of the first dose of study drug.
* Subject has a known sensitivity to any of the components of the investigational product ASP1235 (AGS62P1):

  * ASP1235 (AGS62P1)
  * L-Histidine base
  * L-Histidine HCl
  * α, α -Trehalose Dihydrate
  * Polysorbate 20
* Major surgery within 28 days of the first dose of study drug
* Subject is pregnant or lactating
* Subject has a condition or situation which may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Subject has any medical, psychiatric, addictive or other disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures
* Subject has ocular condition such as:

  * Active infection or corneal ulcer
  * Monocularity
  * History of corneal transplantation
  * Contact lens dependent (if using contact lens, must be able to switch to glasses during the entire study duration)
  * Uncontrolled glaucoma (topical medications allowed)
  * Uncontrolled or active ocular problems (e.g., retinopathy, macular edema, active uveitis, macular degeneration) requiring surgery, laser treatment, or intravitreal injections
  * Papilledema or other active optic nerve disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events | up to 30 months
  AEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) grading scale, version 4.03 (National Institutes of Health, 2010).

SECONDARY OUTCOMES:
Incidence of antidrug antibody (ADA) formation to the fully human monoclonal antibody (AGS62P) and antibody-conjugate (ASP1235 [AGS62P1]) | up to 46 months
Complete response (CR) | up to 46 months
Composite complete remission (CRc) rate | up to 46 months
Best response rate | up to 46 months
Duration of remission | up to 46 months
Duration of response | up to 46 months
Morphologic leukemia free state (MLFS) rate | up to 30 months
Concentration at the end of infusion (CEOI) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Concentration at the end of infusion (CEOI) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Concentration at the end of infusion (CEOI) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Maximum observed concentration (Cmax) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Maximum observed concentration (Cmax) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Maximum observed concentration (Cmax) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Time to maximum concentration (Tmax) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Time to maximum concentration (Tmax) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Time to maximum concentration (Tmax) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Systemic clearance (CL) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Systemic clearance (CL) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Systemic clearance (CL) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Volume of distribution at steady state (Vss) of total antibody (TAb) in dose escalation part | up to an average of 30 months
Volume of distribution at steady state (Vss) of antibody drug conjugate (ADC) in dose escalation part | up to an average of 30 months
Volume of distribution at steady state (Vss) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose escalation part | up to an average of 30 months
Concentration at the end of infusion (CEOI) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Concentration at the end of infusion (CEOI) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Concentration at the end of infusion (CEOI) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Maximum observed concentration (Cmax) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Maximum observed concentration (Cmax) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Maximum observed concentration (Cmax) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Time to maximum concentration (Tmax) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Time to maximum concentration (Tmax) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Time to maximum concentration (Tmax) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Partial area under the serum concentration-time curve (AUC) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Terminal or apparent terminal half-life (t1/2) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Systemic clearance (CL) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Systemic clearance (CL) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Systemic clearance (CL) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months
Volume of distribution at steady state (Vss) of total antibody (TAb) in dose expansion part | up to an average of 30 months
Volume of distribution at steady state (Vss) of antibody drug conjugate (ADC) in dose expansion part | up to an average of 30 months
Volume of distribution at steady state (Vss) of metabolite para-acetyl phenylalanine attached to the microtubule disrupting agent linked to linker 30 (pAF-AGL-0185-30) in dose expansion part | up to an average of 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Officer, Study Director — Astellas Pharma Global Development, Inc.
Locations (7):
- United States (6):
  - Site US00006, Duarte, California
  - Site US00003, Baltimore, Maryland
  - Site US00007, Boston, Massachusetts
  - Site US00009, Boston, Massachusetts
  - Site US00004, New York, New York
  - Site US00001, Houston, Texas
- Site CA00010, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Al Malki MM, Minden MD, Rich ES, Hill JE, Gill SC, Fan A, Fredericks CE, Fathi AT, Abdul-Hay M. Safety, tolerability, and pharmacokinetics of ASP1235 in relapsed or refractory acute myeloid leukemia: A phase 1 study. Leuk Res. 2025 May;152:107690. doi: 10.1016/j.leukres.2025.107690. Epub 2025 Apr 2. PMID 40209615
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=1235-CL-0101/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14552&tenant=MT_AST_9011